CLINICAL TRIAL: NCT06643273
Title: A Multicenter Randomized Controlled Trial on the Effects of Upper Limb Robotic Rehabilitation on Sensory and Cognitive Impairments in Subjects With Stroke. The SCORES (Sensory and Cognitive Outcomes of Robotic Exercises in Stroke) Study. Evaluation of a Haptic Glove.
Brief Title: Evaluation of a Haptic Glove for Assessing Tactile Perception in Post-Stroke Patients
Acronym: SCORES-glove
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCORES-haptic glove; GR-2021-12374896 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: tactile perception; haptic glove; robotics; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Rehabilitation (Experimental): Robotic Rehabilitation of the upper limb
  Interventions: Other: Robotic rehabilitation
- Conventional Rehabilitation (Active Comparator): Conventional Rehabilitation of the upper limb
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Robotic rehabilitation — Upper limb rehabilitation using a set of 4 devices. A set of motor/cognitive exercises will be selected to train also attention, memory, executive function, speed of processing, and visuospatial abilities.The following devices will be used: (a) a robotic device that allows passive, active, and active-assistive planar movements of the shoulder and elbow joints (Motore, Humanware); (b) a robotic device that allows passive, active, and active-assistive finger flexion and extension movements (Amadeo, Tyromotion); (c) a sensor-based system that allows unsupported 3-dimensional movements of shoulder, elbow, and wrist joint, both unimanual and bimanual (Pablo, Tyromotion); and (d) a robotic system that allows 3-dimensional, unimanual and bimanual, movements of the shoulder joint, with arm weight support (Diego, Tyromotion).
  The rehabilitation treatment will be performed daily for 45 minutes, 5 days/week, for a total of 30 sessions.
  Arms: Robotic Rehabilitation
Other: Conventional rehabilitation — Upper limb rehabilitation using conventional techniques, focused on upper limb reprogramming sensorimotor function, hypertonus, inhibition and functional improvement.
  The rehabilitation treatment will be performed daily for 45 minutes, 5 days/week, for a total of 30 sessions.
  Arms: Conventional Rehabilitation

SUMMARY:
The aim of the SCORES Haptic Glove Study is to assess the technical features, safety, and reliability of a sensor-equipped glove designed to evaluate tactile perception. This will help guide further technical and functional improvements to finalize the device. The secondary goal is to validate a new tactile sensitivity index based on data collected using the glove. This will be done in a randomized controlled multicenter study (ClinicalTrials.gov ID NCT06109324) aimed to compare the effectiveness of robotic upper limb rehabilitation to conventional treatment in improving cognitive and sensory deficits, as well as evaluating the impact of these deficits on motor recovery.

DETAILED DESCRIPTION:
Sensory and proprioceptive deficits in the upper limbs affect about 50-85% of stroke survivors. These deficits can impact single sensations (such as primary tactile senses like light touch, pressure, and localization) and the ability to discriminate between different materials or temperatures, as well as proprioception and multiple somatosensory modalities. Furthermore, somatosensory deficits have been strongly correlated with variations in treatment responses among patients. However, in clinical practice, the use of appropriate quantitative tools to measure these deficits is not widespread, and evidence for active sensory training remains limited.

In recent years, robotic therapy has been proposed as an effective approach for upper limb rehabilitation. Nevertheless, recent studies with large samples have failed to demonstrate the superiority of robotic treatment over traditional methods regarding the recovery of upper limb motor functions. These studies primarily focus on motor aspects of stroke recovery, often neglecting sensory and cognitive aspects of rehabilitation, whether robotic or conventional.

Actually, there is limited evidence supporting the superiority of robotic approaches over conventional rehabilitation in recovering cognitive deficits and sensitivity. Additionally, it remains unclear whether cognitive and/or sensory deficits impact motor outcomes differently when using robotic versus conventional approaches.

To address this, the SCORES (Sensory and Cognitive Outcomes of Robotic Exercises in Stroke) study is a multicenter randomized controlled study investigating the effects of robotic rehabilitation on cognitive and sensory deficits in stroke survivors. It aims to compare robotic and conventional rehabilitation approaches regarding cognitive recovery and tactile sensitivity in subacute stroke patients. While some quantitative methods exist to assess absolute perception levels of tactile stimuli, standardized, repeatable, and objectively quantitative methods for assessing localization ability are lacking. Therefore, this study will evaluate how the tactile perceptual abilities of recruited patients evolve during and after a rehabilitation course-whether robotic or conventional-using a specifically developed haptic device that includes a glove with integrated vibrotactile elements. This system aims to objectively define patients' tactile sensitivity through psychophysical evaluations involving the identification and localization of randomized vibrations delivered to the surface of the hand affected by sensorimotor alterations. Specifically, this study will investigate the test-retest reliability, discriminant ability, responsiveness, and clinical validity of the metrics obtained from the haptic glove.

During each experimental session, randomized vibrotactile stimuli will be administered to the recruited patient at different sites on the hand. The patient will be asked to identify and verbally communicate the site of each perceived vibration, as well as the intensity of the vibration itself between the two possible levels.

ELIGIBILITY:
Inclusion Criteria:

* a single event, verified by MRI or CT;
* age between 18 and 85 years;
* time since stroke within six months;
* a demographically adjusted total score of the Montreal Cognitive Assessment (MoCA) between 15.5 and 22.23

Exclusion Criteria:

* behavioural and cognitive disorders and/or reduced compliance that would interfere with active therapy;
* fixed contraction deformity in the affected limb that would interfere with active therapy (ankylosis, Modified Ashworth Scale = 4);
* severe deficits in visual acuity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number and types of the haptic glove malfunctions that occurred during the study, along with their descriptions (Feasibility evaluation) | Baseline; within 2 days after the end of rehabilitation treatment; within 2 days after the end of rehabilitation treatment; 6 months after the end of treatment.
  Number and types of the haptic glove malfunctions that occurred during the study, along with their descriptions.

SECONDARY OUTCOMES:
Number of stimulations provided by the haptic glove and correctly identified in terms of intensity and localization (test-retest reliability) | Baseline; within two day after baseline
  The number of stimulations provided by the haptic glove and correctly identified by the patient in terms of intensity and localization at baseline and within two days after baseline will be assessed to evaluate the measure's test-retest reliability
Number of stimulations correctly identified in terms of intensity and localization (responsiveness) | Baseline; within 2 days after the end of rehabilitation treatment; 6 months after the end of treatment.
  The number of stimulations provided by the haptic glove and correctly identified by the patient in terms of intensity and localization before and after the intervention will be assessed to evaluate the measure's responsiveness
Number of stimulations correctly identified in terms of intensity and localization (clinical validity) | Baseline; within 2 days after the end of rehabilitation treatment.
  The number of stimulations provided by the haptic glove and correctly identified by the patient in terms of intensity and localization before and after the intervention will be correlated with the Semmes-Weinstein monofilament test at the same timepoint to assess measure's clinical validity

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Fondazione Don Carlo Gnocchi, Florence
  - IRCCS Centro Neurolesi Bonino Pulejo, Messina
  - Fondazione Don Carlo Gnocchi - Centro Santa Maria della Provvidenza, Roma

IPD SHARING:
Plan to Share IPD: No